CLINICAL TRIAL: NCT06636370
Title: Contrast-enhanced Mammography and Abbreviated MRI as Supplemental Screening Modalities for Women Aged 50-75 With Extremely Dense Breast Tissue: the DENSE-2 Trial
Brief Title: Supplemental Screening for Women With Extremely Dense Breast Tissue: the DENSE-2 Trial
Acronym: DENSE-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: C.H. van Gils (Other)
Collaborators: University Medical Center Groningen (Other); Ziekenhuisgroep Twente (Other); Radboud University Medical Center (Other); Rijnstate Hospital (Other); Zuyderland Medical Centre (Other); Maastricht University Medical Center (Other); Elisabeth-TweeSteden Ziekenhuis (Other); Catharina Ziekenhuis Eindhoven (Other); Jeroen Bosch Hospital (Unknown); Erasmus Medical Center (Other); Albert Schweitzer Hospital (Other); St. Antonius Hospital (Other); Antoni van Leeuwenhoek Hospital (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Bevolkingsonderzoek Nederland (Unknown); Borstkankervereniging Nederland (Unknown)
Responsible Party: Sponsor-Investigator, C.H. van Gils, Professor Dr., UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 05550412310002; Nr. 2024/09 (Other: Dutch Health Council)
Record Dates: First submitted 2024-10-03; First posted 2024-10-10 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: breast cancer screening; extremely dense breasts; early detection; contrast-enhanced mammography; abbreviated MRI
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): This group receives biennial mammography only within the current Dutch National Breast Cancer Screening program. This group will not be informed about the study (pre-randomisation design)
- Contrast-enhanced Mammography (CEM) (Experimental): This group receives supplemental screening with CEM after a negative mammography result in the Dutch National Breast Cancer screening program
  Interventions: Diagnostic Test: Contrast-enhanced mammography (CEM)
- Abbreviated MRI (AB-MRI) (Experimental): This group receives supplemental screening with AB-MRI after a negative mammography result in the Dutch National Breast Cancer Screening program
  Interventions: Diagnostic Test: Abbreviated MRI (AB-MRI)

INTERVENTIONS:
Diagnostic Test: Contrast-enhanced mammography (CEM) — This intervention group receives supplemental screening with CEM after a negative screening result within the Dutch National Breast Cancer Screening program
  Arms: Contrast-enhanced Mammography (CEM)
Diagnostic Test: Abbreviated MRI (AB-MRI) — This intervention group receives supplemental screening with AB-MRI after a negative screening result within the Dutch National Breast Cancer Screening program
  Arms: Abbreviated MRI (AB-MRI)

SUMMARY:
Women with extremely dense breasts (nearly all glandular and connective tissue, little fatty tissue) have a 3-6 times higher risk of breast cancer than women with very low breast density. Moreover, due to the masking effect of the dense tissue, any breast tumours present are more difficult to detect in these women. With the results of the DENSE trial, the investigators showed that among women with extremely dense breasts, a combination of MRI and mammography could detect tumours earlier than mammography only. As the implementation of MRI in the screening program induces considerable costs and capacity requirements, the Dutch Ministry of Health would like to investigate whether cheaper and acceptable alternatives can be implemented more easily. In the DENSE-2 study, proposed here, we will investigate contrast-enhanced mammography and an abbreviated form of MRI as alternatives, in a large-scale randomized trial, within the current population-based screening program.

DETAILED DESCRIPTION:
Women with extremely dense breast tissue have a higher risk of developing breast cancer and at the same time, mammography has limited value for these women. Currently, these women are not offered supplemental screening. Therefore, the investigators of the DENSE-2 trial will study supplemental CEM and AB-MRI screening in women with extremely dense breast tissue within the population-based breast cancer screening program because these modalities are expected to have higher diagnostic accuracy than tomosynthesis and ultrasound. In addition, these modalities are expected to be less expensive and require less capacity than a full MRI protocol as examined in the DENSE trial. For both CEM and AB-MRI, no results are currently available from a prospective screening study. The DENSE-2 trial is a randomized controlled trial comparing two intervention arms (CEM [intervention arm A] and abbreviated MRI [intervention arm B]) each with mammography [control arm C].

ELIGIBILITY:
Inclusion Criteria:

* Participant in the Dutch population-based breast cancer screening program with a negative mammography result (BI-RADS classification 1 or 2).
* Extremely dense breast tissue (assessed with Quantra software, category D).
* Age between 49-72 years (women are invited to the Dutch screening program in the year they turn 50, so the minimum age is 49 years. The maximum age for inclusion is 72 years to ensure that women can still participate in a second round of supplemental screening).
* Living in the service area (travel distance of up to 60 km) of the 15 participating hospitals.
* Absence of breast implants (Quantra cannot provide an accurate density determination for breasts with implants).
* No objection to data sharing.
* Not a participant in the DENSE trial or STREAM trial (participants in the DENSE and STREAM trials are known to the Dutch screening organization).

Exclusion Criteria:

The additional exclusion criteria for the intervention arms are checked after randomization and recruitment (this order is due to the pre-randomization design):

* Presence of in-body metals (only for AB-MRI, this involves specific metals and is asked by telephone).
* Previous allergic reaction to the provided contrast agent.
* Renal insufficiency (glomerular filtration rate <30 ml/min) (only for CEM, is checked for with questionnaire I and possibly renal function measurement).
* Severe claustrophobia (only for AB-MRI).
* Severe obesity (weight >150 kg) (only for AB-MRI).

Ages: 49 Years to 72 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36000 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Interval Cancer Rate | 0 - 3 year
  Measured as a breast cancer diagnosed in between two screening rounds

SECONDARY OUTCOMES:
Cancer detection rate | 0 - 3 year
  The number of breast cancers detected by CEM or AB-MRI
False positive rate | 0-5 year
  The number with a false positive result after CEM or AB-MRI
Participant experience with CEM - 1 | 0-5 year
  screen-specific item questionnaire (SSI)
Participant experience with CEM - 2 | 0-5 year
  Self-developed questionnaire
Participant experience with CEM - 3 | 0-5 year
  Focus group interviews
Participant experience with AB-MRI - 1 | 0-5 year
  screen-specific item questionnaire (SSI)
Participant experience with AB-MRI - 2 | 0-5 year
  Self-developed questionnaire
Participant experience with AB-MRI - 3 | 0-5 year
  Focus group interviews
Health-professional experience with CEM | 0-5 year
  Self-developed questionnaire
Health-professional experience with AB-MRI | 0-5 year
  Self-developed questionnaire
Estimated rate of overdiagnosis | 0-5 years
  Simulation with the MISCAN software
Cost-effectiveness | 0-5 year
  Simulation with the MISCAN software
Breast tumor size | 0-5 years
  mm
Breast tumor stage | 0-5 years
  TNM classification
Positive Predictive Value (PPV) | 0-5 year
  Using the histological diagnosis as the reference test
Biopsy rate | 0-5 year
  Per 1000 women screened with one of the modalities
Referral rate | 0-5 years
  Per 1000 women screened per screening modality
Mortality rate | 0-5 year
  Simulation with MISCAN software

CONTACTS AND LOCATIONS:
Overall Officials: Carla van Gils, Prof., Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided